CLINICAL TRIAL: NCT05544253
Title: Safety and Efficacy of Mitomycin C-based Hyperthermic Intraperitoneal Chemotherapy After Spontaneously Ruptured Hepatocellular Carcinoma and Peritoneal Metastasis: a Randomized Controlled Trial
Brief Title: Safety and Efficacy of Mitomycin C-based HIPEC After srHCC and PM of HCC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiwei Huang, Department of Liver Surgery and Liver Transplantation Centre, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHuang
Record Dates: First submitted 2022-09-10; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma; Peritoneal Metastasis; Hyperthymic; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIPEC group (Experimental)
  Interventions: Procedure: mitomycin C-based hyperthermic intraperitoneal chemotherapy
- non-HIPEC group (No Intervention)

INTERVENTIONS:
Procedure: mitomycin C-based hyperthermic intraperitoneal chemotherapy — The patients with srHCC or PM of HCC were randomly allocated to either the HIPEC group or the control group. All of them have received open liver resection and perfusion tubes had been set in the operation. For patients with PM of HCC served operation, we are subject to reach CC score at 0-1 to creating sufficient conditions for HIPEC. Finally, place the HIPEC tubes. Implementation of HIPEC was administered 3times on the 1st, 3rd, 5th days within one week after operation. We used intraperitoneal hyperthermic perfusion device (BR-TRG-IITM, Bao Rui medical corporation, Guangdong, China) to achieve HIPEC. The abdominal temperature was maintained at 43°C (109°F) by circulating heated saline. The perfusion volume was 3000ml of normal saline, and the chemotherapeutic agent of mitomycin C was 10mg for a 1-hour perfusion period.
  Arms: HIPEC group

SUMMARY:
Hepatocellular carcinoma (HCC) is featured by the spontaneously rupture when suffering severe cirrhosis and intratumoral overpressure. It is a fatal complication with an acute mortality. Importantly, it is served as an independent risk factor for peritoneal metastasis (PM) of HCC with poor prognosis. The systematic agents effective to extrahepatic lesions confers modest efficacy towards PM. HIPEC, as a novel strategy, has been proved by overwhelming studies that it is effective to peritoneal malignant tumors. However, there is absence of prospective study of HIPEC efficacy towards HCC.

ELIGIBILITY:
Inclusion Criteria:

1. HCC patients have been diagnosed by NCCN clinical practice guidelines in oncology, Hepatobiliary cancers, version 2.2021.
2. ECOG score of 0-2 points;
3. Child-Pugh class A-B liver function only;
4. Consistent with the diagnosis of srHCC: symptoms: acute abdominal pain and peritonitis; blood routine tests: decrease of erythrocyte count; increase of leucocyte count, especially the proportion of neutrophils; radiological features: contrast materials extravasation from lesions confirmed by abdominal contrast enhanced computed tomography or promethean magnetic resonance imaging; intraoperative findings of tumor rupture and postoperative pathology are more confidently conclusive.
5. Consistent with PM of HCC: histological evaluations: biopsy of peritoneal nodules or ascites cytology or postoperative pathological verification; radiological diagnose: early enhancement and late wash-out radiological property of peritoneal nodule or mutual confirmation by two senior radiologists.
6. All of selections have received open or laparoscopic hepatectomy to reach complete macroscopic resection or less than 2.5mm of residual tumor tissue, which is equal to 0 or 1 degree of completeness of cytoreduction.
7. Patients voluntarily participated and signed the informed consent.

Exclusion Criteria:

1. Contraindications of HIPEC, such as: extensive intra-abdominal adhesions caused by various reasons; complete intestinal obstruction; severe kidney insufficiency; myelosuppression caused by previous targeted therapy or own blood system disease; severe cardiovascular system disease; infection, especially abdominal infection; bleeding tendency or coagulation dysfunction; the vital signs are unstable; cachexia;
2. Extraperitoneal metastasis;
3. Patients who refuse to accept clinical trials;
4. Those who are deemed unsuitable for inclusion by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
recurrence-free-survival | 2years
  the time from the first administration to the date of first recurrence, including local recurrence and PM and distant metastasis, or death for any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No